CLINICAL TRIAL: NCT04842942
Title: The Safety and Feasibility of Transoral Endoscopic Thyroidectomy Vestibular Approach
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-5679
Record Dates: First submitted 2021-02-19; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Thyroid Diseases; Surgery
Keywords: TOETVA; Transoral Endoscopic Thyroidectomy Vestibular Approach
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Intervention Model Description: The study intervention in this study is the TOETVA-procedure. This is an Transoral Endoscopic Thyroidectomy Vestibular Approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOETVA (Experimental): Transoral Endoscopic Thyroidectomy Vestibular Approach
  Interventions: Procedure: TOETVA

INTERVENTIONS:
Procedure: TOETVA — Transoral Endoscopic Thyroidectomy Vestibular Approach

SUMMARY:
This is a single center, prospective case series designed to assess the safety and feasibility of TOETVA in a small cohort of patients at University Health Network Toronto. Included patients will undergo a TOETVA-procedure in stead of the standard open surgical procedure.

DETAILED DESCRIPTION:
Type of Study This is a single center, prospective case series

Sample Size Since this is a feasibility study we will first include 15 patients. If we find the TOETVA a safe and feasible approach, we will perform the same study in more patients using the results of this study for a power size calculation.

Study Population Patients (> 18 years) undergoing (para)thyroid surgery for the indication of a benign or indeterminate thyroid nodule, well differentiated papillary thyroid carcinoma, well-controlled Grave's disease or a parathyroid adenoma.

Study Design This is a single center, prospective case series designed to assess the safety and feasibility of TOETVA in a small cohort of patients at University Health Network Toronto. Included patients will undergo a TOETVA-procedure in stead of the standard open surgical procedure.

Study Intervention The study intervention in this study is the TOETVA-procedure. This is an Transoral Endoscopic Thyroidectomy Vestibular Approach.

Primary Objective The study objective is to assess the safety and feasibility of this procedure in a small cohort of patients at University Health Network Toronto, Ontario.

Endpoints of the study The main study endpoints consist of

1. Surgical Outcomes: rate of post-operative recurrent laryngeal nerve palsy, rate of post-operative hypocalcemia, and rate of neck incision (conversion to open), oral infections, neck infection, hematoma, seroma, subcutaneous emphysema, gas-induced embolism, surgical time, and length of stay.
2. Quality of Life - EORTC Thyroid specific Health related quality of life

These endpoints will be compared to historical age/indication controls for analysis.

ELIGIBILITY:
Inclusion Criteria:

- Patients needing surgery for: Benign or indeterminate nodule less than 6 cm in size or; T1 well differentiated papillary carcinoma less than 2 cm in size or; Well-controlled Grave's disease or; Parathyroid adenoma.

* Total thyroid size is 7-8 cm (no more than 10 cm)
* Their age is ≥18 years and ≤80 years
* Able to give written consent

Exclusion Criteria:

* - History of neck surgery or neck radiotherapy
* Recurrent thyroid disease
* Lymph node metastases
* Presence of intraoral infections
* Presence of extrathyroidal or substernal extensions
* Smoking
* Morbid obesity
* Contra-indication to general anesthesia with nasotracheal intubation
* Previous mediastinal surgery
* Any anatomical anomaly that in the opinion of the investigator may render the intervention more difficult (ex. variations in the structure of the platysmas muscle)
* Any medical condition, which in the judgment of the investigator and/or designee makes the subject a poor candidate for the investigational procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Post-operative recurrent laryngeal nerve palsy | 12 months
  Number of participants with post-operative recurrent laryngeal nerve palsy
Postoperative hypocalcemia | 12 months
  Number of participants with postoperative hypocalcemia
Neck incision | 1 month
  Number of conversions to open
Rate of oral infections | 12 months
  Number of participants with oral infections
Rate of hematoma | 1 month
  Number of participants with hematomas
Rate of seroma | 1 month
  Number of participants with seromas
Rate of neck infection | 12 months
  Number of participants with neck infections
Rate of subcutaneous emphysema | 12 months
  Number of participants with subcutaneous emphysema
Rate of gas-induced embolism | 12 months
  Number of participants with gas-induced embolism
Surgical time | until surgical discharge, average of 24 hours
  Surgical time in hours
Length of stay | until surgical discharge, average of 24 hours
  Length of stay in days

SECONDARY OUTCOMES:
Quality of Life Score | 12 months
  EORTC Thyroid specific Health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jesse D Pasternak, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Univeristy Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No